CLINICAL TRIAL: NCT01762176
Title: Effect of Early Intensive Treatment in Chinese Patients With Recent-onset Rheumatoid Arthritis
Brief Title: Early RA MRI Early Intensive Treatment Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Lai-Shan Tam, Professor, Chinese University of Hong Kong
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ERA-MRI-2012
Record Dates: First submitted 2013-01-04; First posted 2013-01-07 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-09

CONDITIONS: Early Rheumatoid Arthritis
Keywords: Early Rheumatoid Arthritis; Usual care; Intensive Care; Boolean criteria
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care group (Active Comparator): Usual care
  Interventions: Procedure: Usual care
- Intensive care group (Active Comparator): Protocolized intensive treatment
  Interventions: Procedure: Protocolized intensive treatment

INTERVENTIONS:
Procedure: Protocolized intensive treatment — Intensive treatment is defined as early diagnosis, frequent assessment (monthly) of disease activity that guides treatment change with the aim to achieve clinical remission based on a tight control protocol
  Arms: Intensive care group
Procedure: Usual care — Usual care is defined as treatment decision at the discretion of the rheumatologists and patients reflecting daily clinical practice
  Arms: Usual care group

SUMMARY:
To compare the effectiveness of two treatment strategies in early rheumatoid arthritis (ERA), namely the delayed usual care and early intensive care, in Hong Kong.

* The delayed usual care reflects the usual treatment practice in Hong Kong
* The early intensive care includes tight monitoring and immediate adjustment of therapy

DETAILED DESCRIPTION:
This study is a 1-year non-randomized clinical trial. Two groups of patients (delayed usual care and early intensive care) with diagnosis of rheumatoid arthritis (RA) and with symptoms onset of less than 2 years and disease modifying anti-rheumatic drugs (DMARDs) naive will be recruited. Remission is reached if patients fulfill the Boolean criteria.

ELIGIBILITY:
Inclusion Criteria:

For usual care group:

* patients with at least 1 tender and swollen joint
* duration of symptoms less than 2 years
* no previous use of DMARDs

For intensive care group:

* patients with at least 1 tender and swollen joint
* duration of symptoms less than 2 years
* no previous use of DMARDs
* patients who fulfill the 2010 ACR/EULAR classification criteria for RA

Exclusion Criteria:

* patients with renal impairment (on dialysis or estimated Glomerular Filtration Rate (eGFR) <30 mL/min/1.73m^2)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2012-10; Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who achieve clinical remission | 12 months
  The clinical remission is defined using the latest ACR/EULAR remission criteria (Boolean criteria)

SECONDARY OUTCOMES:
Change in various patient-reported outcomes | 12 months
  The various patient-reported outcomes include employment status, Working Ability Index (WAI), disability index of Health Assessment Questionnaire (HAQ), Functional Assessment of Chronic Illness Therapy (FACIT), Hospital Anxiety and Depression Scale (HADS) and Health-related quality of life (HRQoL) generic measures
Gains in utility | 12 months
  The Utility score is calculated by EQ-5D self-report questionnaire, which provides a single index value for health status that can be used in the clinical and economic appraisal. Value set derived from a Chinese cohort in Beijing is used, since no value set for Hong Kong Chinese population is available.
Radiographic progression | 12 months
  Radiographic progression expressed using the van der Hejide modification of the Sharp scored
ACR 20, 50, 70 responses | 12 months
  The ACR 20, 50, 70 responses are defined as at least 20%, 50%, 70% improvement in joint swelling and joint tenderness counts, and at least three of five other variables (i.e. erythrocyte sedimentation rate, HAQ score, pain score, and physicians' and patients' global assessments)
MRI outcome | 12 months
  MRI image set is evaluated and scored separately for the presence or absence of MRI erosion, synovitis, and bone marrow oedema. Bone erosions and bone marrow oedema are evaluated separately in each wrist bone, whereas synovitis is evaluated in the three regions of the wrist joint: the radioulnar area, the radiocarpal area, and the intercarpal-carpometacarpal area.

CONTACTS AND LOCATIONS:
Overall Officials: Lai Shan Tam, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, China